CLINICAL TRIAL: NCT07101055
Title: A Prospective, Open-Label, Single-Centre, Comparative Pharmacokinetic Study of Oral Letermovir (PREVYMIS) in Patients (i) Undergoing Intermittent Haemodialysis and (ii) Not Undergoing Intermittent Haemodialysis
Brief Title: Pharmacokinetics of Oral Letermovir in Adults With End-Stage Kidney Disease With or Without Haemodialysis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jason A Roberts (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Royal Brisbane and Women's Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Jason A Roberts, Professor, The University of Queensland
Organization: The University of Queensland (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UQ117254-Letermovir
Record Dates: First submitted 2025-07-22; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: End-Stage Kidney Disease (ESKD)
Keywords: pharmacokinetics; letermovir; intermittent haemodialysis; renal impairment; chronic kidney failure
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency | interventions — letermovir

STUDY DESIGN:
Intervention Model Description: Participants are enrolled into two parallel groups based on dialysis status: adults with end-stage kidney disease (i) undergoing intermittent haemodialysis, and (ii) not undergoing dialysis. Each participant receives a single oral dose of letermovir (480 mg), and pharmacokinetic profiles are compared between groups. There is no randomisation or crossover.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESKD undergoing intermittent haemodialysis (Experimental): Participants with end-stage kidney disease (ESKD) who are receiving regular intermittent haemodialysis. Each participant receives a single oral dose of letermovir (480 mg) approximately 2 hours before their scheduled dialysis session.
  Interventions: Drug: Letermovir 480 mg [PREVYMIS]
- ESKD not undergoing intermittent haemodialysis (Experimental): Participants with end-stage kidney disease (ESKD) who are not receiving haemodialysis. Each participant receives a single oral dose of letermovir (480 mg).
  Interventions: Drug: Letermovir 480 mg [PREVYMIS]

INTERVENTIONS:
Drug: Letermovir 480 mg [PREVYMIS] — A single 480 mg oral dose of letermovir (2 x 240 mg tablets).

SUMMARY:
This study aims to understand how the antiviral medication letermovir (PREVYMIS) is processed by the body in adults with end-stage kidney disease (ESKD), including those who are receiving intermittent haemodialysis and those who are not. Letermovir is already approved in many countries, including Australia, for preventing cytomegalovirus (CMV) infections in patients who have received stem cell transplants. However, its pharmacokinetics - or how the drug is absorbed, distributed, and cleared from the body - have not been studied in patients with ESKD, especially those on dialysis.

This is a single-centre, open-label, interventional pharmacokinetic study. It will recruit 20 adult participants, split into two groups: 10 participants on intermittent haemodialysis and 10 not undergoing dialysis. All participants will receive a single oral dose of 480 mg letermovir. The study does not involve treatment for CMV infection. Instead, it focuses only on how the drug behaves in the body in this patient population.

Participants will have blood samples collected before and after taking the medication to measure drug concentrations over time. In patients on dialysis, an additional sample will be taken from the dialysis machine to understand if letermovir is removed during treatment. No more than 35 mL of blood (around two tablespoons) will be collected across two study visits.

The goal of this study is to generate important safety and dosing information to help guide future use of letermovir in people with kidney failure. It is expected that these findings will support more informed clinical decisions and potentially lead to updated dosing recommendations for this group.

The study is funded by Merck Sharp & Dohme LLC (MSD), the manufacturer of letermovir, and is being conducted by researchers from The University of Queensland Centre for Clinical Research (UQCCR) and the Royal Brisbane and Women's Hospital (RBWH). To support participation, prepaid meal vouchers, taxi vouchers, or parking tickets will be provided so that participants do not incur any out-of-pocket expenses.

Participation is voluntary. The study has been approved by a Human Research Ethics Committee and is conducted according to national ethical guidelines.

ELIGIBILITY:
Inclusion Criteria:

All participants of childbearing potential who are engaging in sexual activity that could result in pregnancy must be willing to use highly effective contraception from screening through 30 days post-dose of letermovir. Male participants must also agree not to donate sperm during this period.

Group 1:

* Adult participants (≥18 years old).
* Estimated Glomerular filtration rate (eGFR) < 15 mL/min/1.73 m2.
* Clinical indication for regular intermittent haemodialysis.
* Agreement to receive a single 480 mg dose of letermovir.
* Willing and able to provide informed consent.
* Consent to cannula placement for blood draws.

Group 2:

* Adult participants (≥18 years old).
* Estimated Glomerular filtration rate (eGFR) < 15 mL/min/1.73 m2.
* No clinical indication for regular intermittent haemodialysis.
* Agreement to receive a single 480 mg dose of letermovir.
* Willing and able to provide informed consent.
* Consent to cannula placement for blood draws.

Exclusion Criteria:

* Participants who lack the capacity to provide informed consent.
* Patients with suspected or known hypersensitivity to any of the active or inactive ingredients of the oral letermovir formulation.
* Patients who are taking any of the following medications, unless these can be safely discontinued temporarily for the duration of the study as determined by the study investigator: statins (pitavastatin, simvastatin, atorvastatin, fluvastatin, lovastatin, pravastatin, rosuvastatin) and proton pump inhibitors (omeprazole, pantoprazole).
* Patients who are taking any of the following medications: cyclosporine, pimozide, ergot alkaloids, or drug metabolism inducers including amiodarone, nafcillin, warfarin, carbamazepine, phenobarbital, phenytoin, glyburide, voriconazole, rifabutin, rifampicin, pimozide, thioridazine, bosentan, St. John's Wort, efavirenz, etravirine, nevirapine, sirolimus, tacrolimus, modafinil, CYP2C8 substrates (e.g., repaglinide, rosiglitazone), or CYP3A substrates (e.g., alfentanil, fentanyl, midazolam, quinidine).
* Patients with severe hepatic impairment.
* Pregnant, planning to conceive, breastfeeding, or intending to breastfeed during the study period.
* Presence of any rapidly progressing disease or immediately life-threatening illness (i.e., death deemed imminent within 48 hours).
* Any condition or circumstance that, in the investigator's opinion, would compromise patient safety or the integrity of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Area Under the plasma concentration-time Curve (AUC) of letermovir | Pre-dose to 48 hours post-dose
  The AUC will be calculated using non-compartmental analysis based on serial plasma concentration measurements following a single oral dose of letermovir. The aim is to compare systemic exposure between participants with end-stage kidney disease who are undergoing intermittent haemodialysis and those who are not.

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Roberts, PhD, Principal Investigator — The University of Queensland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the small sample size and the potential for re-identification of participants with end-stage kidney disease, a vulnerable population. In addition, IPD sharing is not covered under the current ethics approval or participant consent.